CLINICAL TRIAL: NCT06882304
Title: PREVALENCE OF WHITE SPOT LESIONS IN ENAMEL AFTER ORTHODONTIC
Brief Title: PREVALENCE OF WHITE SPOT LESIONS IN ENAMEL AFTER ORTHODONTIC TREATMENT IN YOUNG ADULTS
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AYATELLAH MOHAMED OSMAN MOHAMED MOHAMED GHONIMA, Ayatellah Mohamed, Cairo University
Other Study IDs: WSL
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: White Spot Lesion
MeSH Terms: interventions — Orthodontics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: orthodontic treatment — young adult after orthodontic treatment

SUMMARY:
The aim of the study is to measure prevalence of enamel white spot lesions in enamel in young adults after orthodontic treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients whose age between 18-30 years old consulting in the outpatient clinic.
2. Provide informed consent.
3. Co-operative patients approving to participate in the trial.
4. Both sexes are included
5. Egyptian -

Exclusion Criteria:

1. Patients under or over this age group.
2. Patients with other developmental defect, such as; fluorosis, amelogenesis imperfecta and syndromes associated with enamel formation defects.
3. Patient with MIH .
4. Refuse to participate in the study.

Ages: 18 Years to 30 Years | Sex: All
Age Groups: Adult
Study Population: 1. Patients whose age between 18-30 years old consulting in the outpatient clinic.
  2. Provide informed consent.
  3. Co-operative patients approving to participate in the trial.
  4. Both sexes are included
  5. Egyptian
Sampling Method: Non-Probability Sample
Enrollment: 368 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of white spot lesions in enamel after orthodontic treatment in young adults | baseline
  to measure the prevalence of enamel white spot lesions in enamel in young adults after orthodontic treatment.

REFERENCES:
- [Background] Tufekci E, Dixon JS, Gunsolley JC, Lindauer SJ. Prevalence of white spot lesions during orthodontic treatment with fixed appliances. Angle Orthod. 2011 Mar;81(2):206-10. doi: 10.2319/051710-262.1. PMID 21208070
- [Background] Akin M, Tezcan M, Ileri Z, Ayhan F. Incidence of white spot lesions among patients treated with self- and conventional ligation systems. Clin Oral Investig. 2015 Jul;19(6):1501-6. doi: 10.1007/s00784-014-1382-3. Epub 2014 Dec 13. PMID 25502686